CLINICAL TRIAL: NCT02551562
Title: A Post-market, Randomized Study to Assess the Efficacy of Skin Rejuvenation Therapy in Combination With Neurotoxin and Full Facial Filler Treatments
Brief Title: A Study to Assess the Efficacy of Skin Rejuvenation Therapy in Combination With Neurotoxin and Full Facial Filler Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DeNova Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NuD-SD-01
Record Dates: First submitted 2015-09-14; First posted 2015-09-16 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Subjects Requesting and Requiring Facial Rejuvenation With Neurotoxins and/or Hyaluronic Acid Fillers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Basic Skin Care (Placebo Comparator): Subjects will use a basic skin care regime following a full facial rejuvenation with hyaluronic acid soft-tissue filler and botulinum neurotoxin.
  Interventions: Other: Placebo
- Group B: NuDerm® System (Experimental): Subjects will use the Nu-Derm® system following a full facial rejuvenation with hyaluronic acid soft-tissue filler and botulinum neurotoxin.
  Interventions: Other: NuDerm® System

INTERVENTIONS:
Other: NuDerm® System — The Nu-Derm® System (Valeant Pharmaceuticals North America, LLP) is a skin care system that helps correct and reduce visible signs of aging such as age spots, rough skin, erythema, sallowness, and hyperpigmentation.
  Arms: Group B: NuDerm® System
Other: Placebo — Basic skin care regimen
  Arms: Group A: Basic Skin Care

SUMMARY:
20 female subjects, between the ages of 25 and 60, who request a full facial rejuvenation treatment, meet all the inclusion and none of the exclusion criteria, and have signed a written informed consent, will be enrolled. Subjects will be divided randomly into two treatment groups:

1. Group A: subjects will use a basic skin care regime following a full facial rejuvenation with hyaluronic acid soft-tissue filler and botulinum neurotoxin.
2. Group B: subjects will use the Nu-Derm® system following a full facial rejuvenation with hyaluronic acid soft-tissue filler and botulinum neurotoxin.

The study consists of 5 visits: Baseline/Screening Assessments (Visit 1), Treatment (Visit 2), Two-Week Evaluation (Visit 3), Six-Week Evaluation (Visit 4), and Twelve-Week Evaluation (Visit 5).

Changes in the subjects' quality of skin will be determined by the PI's assessment of skin tone (dyschromia), elasticity (firmness), texture (smoothness), radiance, and wrinkling as well as the global aesthetic improvement at 6 and 12 weeks following neurotoxin and hyaluronic acid treatments. The PI will be blind to the group assignment of the subjects.

Subjects' satisfaction with treatments and their quality of skin will be determined through a self-evaluation at 6 and 12 weeks following neurotoxin and hyaluronic acid treatments. The impact of treatments on subjects' state self-esteem will also be assessed at 6 and 12 weeks following the treatments.

ELIGIBILITY:
Inclusion Criteria:

* Subject requires a full facial rejuvenation with a HA soft tissue filler and/or botulinum neurotoxin, per judgment of the PI;
* Subject is willing and able to provide written informed consent prior to the performance of any study related procedure;
* Subject is willing and able to comply with the protocol requirements; and
* Subject is willing and able to provide written photo consent and adhere to the photography and video procedures such as removal of jewelry and makeup.

Exclusion Criteria:

* Subjects who have received any facial filler or neurotoxin treatments in the 12-month period prior to enrollment;
* Previous treatment with any facial aesthetic procedure (e.g. chemical peeling, photo rejuvenation, and laser treatments) within the 12-month period prior to enrollment;
* Subjects who plan to undergo facial cosmetic surgery or any aesthetic procedure (e.g. neurotoxins, dermal fillers, laser treatments, and chemical peels), which are not specified in this protocol, during the course of the study;
* A known allergy or sensitivity to any component of the study ingredients;
* Use of systemic steroids or anticoagulation medications;
* Subjects with a history of bleeding disorders;
* Subjects with severe allergies manifested by a history of anaphylaxis or presence of multiple severe allergies;
* Subjects with hypersensitivity to botulinum neurotoxin;
* Subject with allergies to gram positive bacterial proteins;
* Sensitivity to sulfides;
* Subjects with allergy to cow's milk protein;
* Subjects with previous history of sensitivity to amide type local anesthetics;
* Subject with surgical alterations to the facial anatomy or marked facial asymmetry;
* Inflammation or infection at the injection site(s);
* Subjects with a history of eyelid or eyebrow ptosis;
* Excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin;
* Subjects with neuromuscular disorders;
* Use of anticholinergic, aminoglycosides or other agents that interfere with neuromuscular transmission (e.g., curare-like agents), or muscle relaxants;
* Subjects with immunodeficiencies such as HIV, lupus, scleroderma, and systemic infections;
* Pregnant, nursing, or sexually active female subjects who are of childbearing potential and who are not willing to use an acceptable form of contraception (e.g., barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence);
* Current history of chronic drug or alcohol abuse;
* Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study product;
* Subjects who, in the investigator's opinion, have a history of poor cooperation, non-compliance with medical treatment, or unreliability; and
* Enrollment in any active study involving the use of investigational devices or drugs.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10-06 (Actual); Primary Completion 2016-09-09 (Actual); Study Completion 2016-09-09 (Actual)

PRIMARY OUTCOMES:
Overall aesthetic improvements | 90 Days
  The primary objective of this study is to examine the effect of skin rejuvenation therapy in combination with full facial rejuvenation, via neurotoxin or HA soft-tissue filler, on the overall aesthetic improvements.

SECONDARY OUTCOMES:
State Self-Esteem | 90 Days
  The secondary objective of this study is to assess the impact of skin quality and aesthetic improvements on short-term self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Dayan, MD, Principal Investigator — DeNova Research
Locations (1):
- DeNova research, Chicago, Illinois, United States